CLINICAL TRIAL: NCT04111016
Title: Exploring the Feasibility of Implementing an Integrated Nutrition, Early Childhood Development and WASH (RINEW) Intervention Through the Government Health System: A Pilot Study
Brief Title: Feasibility of Implementing RINEW Through the Government System
Acronym: RINEW
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); University of California, Berkeley (Other); Johns Hopkins University (Other); BRAC University (Other)
Responsible Party: Principal Investigator, Stephen P Luby, Professor of Medicine (Infectious Diseases), Stanford University
Other Study IDs: 50733
Record Dates: First submitted 2019-05-30; First posted 2019-10-01 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Early Childhood Development
Keywords: Early childhood development; Responsive parenting; Nutrition; WASH; Stimulation; Parenting; Integrated Interventions
MeSH Terms: interventions — Nutritional Status; Lead; Arsenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants able to access the intervention: These group sessions will be delivered by government health workers, and include behavioral recommendations about responsive stimulation, nutrition, water, sanitation and hygiene, lead poisoning prevention, and maternal mental health. Pregnancy groups and caregiver-child groups will be held separately, and mothers and caregivers who attend sessions will receive simple toys and books to use during some of the intervention sessions, which they will be permitted to take home with them. In addition, mothers and caregivers who attend intervention sessions will receive 30 sachets containing 1 gm multiple micronutrient powder (MNP) per month. Beginning as soon as pregnancy is confirmed, health workers will facilitate pregnant women in receiving the Iron and Folic acid supplements already provided by the Government of Bangladesh and will continue the supplementation up to three months post-partum period.
  Interventions: Behavioral: Integrated child stimulation, nutrition, lead, arsenic, WASH intervention

INTERVENTIONS:
Behavioral: Integrated child stimulation, nutrition, lead, arsenic, WASH intervention — The content of the intervention curriculum was developed considering the needs of the specific ages of the children attending the group, as well as the feasibility of delivering the package in the community. The pregnancy module encompasses information on significance of prenatal care for child development, physiological symptoms and solutions, maternal diet, education on kangaroo mother care (KMC), breast feeding, thinking healthy, hygiene, and lead and arsenic prevention. The curriculum for lactating mothers focuses on specialized messages for 4 age groups of children: 0-5 months, 6-11 months, 12-18 months and 19-24 months. The overall package includes information regarding WASH, psychosocial stimulation, nutrition, maternal mental health, lead and arsenic. As research evidence showed that psychosocial stimulation provided for 10 or 12 months can significantly improve child development, the psychosocial stimulation component is included in every fortnightly session.

SUMMARY:
The goal of this study is to assess the feasibility of implementing a group-based integrated early child development intervention through the government health system in one sub-district of Bangladesh, and to assess the resulting uptake of the intervention in the target population.

DETAILED DESCRIPTION:
The RINEW intervention is a group-based integrated nutrition, responsive stimulation, and WASH intervention with a goal to improve child development outcomes. The intervention is delivered in group sessions to pregnant women and mothers or primary caregivers of children under 24 months of age. The RINEW intervention was tested in a pilot cluster-randomized control study in Bangladesh, where the investigators found the intervention group had better self-reported knowledge and behavior related to early child development. The investigators aim to implement this intervention through the government health system in one sub-district of Bangladesh, and assess the feasibility of delivering the intervention in this way, as well as the uptake of the intervention in the target population. The facilitators will be trained by the study team, and the intervention will be implemented in community-level health centers, facilitated by government health workers.

The specific objectives of this work are to:

1. Assess the feasibility (i.e. satisfaction of providers, perceived appropriateness of content and practicability of session delivery, population demand for sessions, quality and frequency of implementation, and preparedness of health system) of implementing the RINEW intervention through the government health system
2. Identify barriers, facilitators/opportunities, and pathway for scale up of the RINEW intervention through government health system
3. Assess the coverage of the intervention in the target population
4. Assess the uptake of recommended behaviors in the target population

To reach these objectives the investigators will

1. Train government health workers to deliver the intervention at government health facilities
2. Conduct a clinic-based process evaluation using both quantitative and qualitative methods at multiple time points during the 12-months intervention
3. Conduct population-based quantitative baseline and endline assessments to assess intervention coverage and uptake

ELIGIBILITY:
Inclusion criteria for household assessment of study participants:

1. mother or primary caregiver of a child 6-24 months old,
2. living in Chatmohar sub-district
3. planning to reside in that area for at least one year (Baseline), or
4. having lived in the area for at least 1 year (Endline).

Exclusion criteria for household assessment of study participants:

1) Child, mother, or primary caregiver with impaired cognitive development, or hearing, vision, speech impaired child or mother.

Inclusion criteria for interviews with study facilitators

1) Government health workers who are participating in the facilitation or supervision of RINEW sessions

Inclusion criteria for qualitative interviews with intervention attendees 1) Mothers or primary caregivers eligible for the intervention sessions

Exclusion criteria for qualitative interviews with intervention attendees

1) Child, mother, or primary caregiver with impaired cognitive development, or hearing, vision, speech impaired child or mother

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chatmohar sub-district of Pabna has been selected to implement the integrated intervention through the government system. All Chatmahor residents with children <2 or families of pregnant women are eligible to participate (attend health facilities offering the intervention)
  The selection of Chatmohar was based on meeting the following criteria:
  i. Communication status from Dhaka: should have a good by road communication (Bus/train) ii. Presence of a local champion in the government health system: UH&FPO should be known and enthusiastic to implement an integrated intervention in the sub-district iii. Low percentage of vacant posts for government frontline health workers: <25% vacant posts iv. Most of the community clinic should be active v. Receptive and less conservative community vi. Community that is exposed to arsenic and lead contamination
Sampling Method: Non-Probability Sample
Enrollment: 2823 (Actual)
Dates: Start 2019-04-06 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Change in session quality | 2nd, 6th and 12th month of the intervention; ~60 min per assessment
  Semi-structured checklist for one pregnancy session and one mother-baby session in each health facility per assessment time period.
Change in proportion of planned session conducted | Every 2 weeks through study completion; ~10 min
  This data will be reported by the intervention facilitators and collected by the intervention supervisors on a monthly basis.
Change in number and proportion of eligible pregnant women and mother attendees at each session | Monthly through study completion; ~15 min/assessment
  The attendance numbers will be collected at each pregnancy and mother-baby session, and reported to the study team on a monthly basis.
Change in satisfaction of trained health workers with training and intervention implementation: Semi-structured individual interviews and focus group discussions | 2nd, 6th and 12th month of the intervention; ~20 min per assessment
  Semi-structured individual interviews and focus group discussions with intervention implementors and their supervisors.
Change in determinants of session quality | 2nd, 6th and 12th month of the intervention; ~20 min per assessment
  Semi-structure individual interviews and focus group discussions with a purposive sample of intervention implementors, their supervisors, and intervention attendees
Change in determinants of session attendance | 2nd, 6th and 12th month of the intervention; ~20 min per assessment
  Semi-structure individual interviews and focus group discussions with a purposive sample of intervention implementors, their supervisors, and intervention attendees

SECONDARY OUTCOMES:
Change in individual-level attendance records and self-reports | Monthly through study completion; ~3 min/assessment
  Attendance to group sessions over the intervention period will be recorded on participant-held attendance records. At the end line assessment participants will also be asked to show their intervention cards and report the number of sessions they have attended over the previous 12 months.
Change in caregiver early child development knowledge and practices | Baseline and 12 months after intervention; ~15 min/assessment
  A modified version of the Family Care Indicators (FCI), including self-reported behaviors and knowledge and observations during the interview, will be used to measure childhood development knowledge and practices. The FCI has the following sub-scales: 1) household books (number); 2) magazines or newspapers in the household (number), 3) sources of play materials (number of 3 possible categories), 4) varieties of play materials (number of 7 possible categories), 5) play activities (number of 6 possible categories). The scores from each sub-scale are summed to calculate the total score. For all sub-scales and the total score, higher scores are associated with a better child care. Investigators will also assess 11 additional observational items including observations of the home environment, and parental responsiveness and acceptance during the interview. Positive responses are summed to create an observation score.
Change in child dietary diversity, child minimum meal frequency and minimum acceptable diet. | Baseline and 12 months after intervention; ~15 min/assessment
  Child dietary diversity will be calculated based on the number of 7 different food groups consumed by the child yesterday. This will be determined based on a maternal-reported 24 hour recall of all foods consumed by the mother and the child. Minimum acceptable diet is determined by the child's dietary diversity and meal frequency.
Change in maternal dietary diversity | Baseline and 12 months after intervention; ~5 min/assessment
  Maternal dietary diversity indicated by the number of 10 different food groups consumed by the mother yesterday. This will be determined based on a maternal-reported 24 hour recall of all foods consumed by the mother and the child.
Change in maternal depressive symptoms | Baseline and 12 months after intervention; ~5 min/assessment
  Caregiver mental health will be measured using the Center for Epidemiologic Studies Depression scale (CESD), which includes 20 questions about symptoms experienced in the previous week. Number of days experiencing each symptom in the last week is converted into a score: 0= 0 or less than 1 day; 1= 1-2 days; 2= 3-4 days, 3=5-7 days, and the total score is a sum of negative symptoms experienced (positive items are reverse scored). The score ranges from 0-60, with higher scores indicating more depressive symptoms experienced.
Change in maternal knowledge regarding lead, nutrition, WASH, and arsenic | Baseline and 12 months after intervention; ~5 min/assessment
  This will be assessed with self-report questions about knowledge about lead exposure and prevention, nutrition, WASH, and arsenic exposure.
Change in self-reported behaviour regarding prevention of lead contamination, disposal of human and chicken feces, water and food storage | Baseline and 12 months after intervention; ~5 min/assessment
  This will be assessed with self-reported questions about behaviours regarding prevention of lead contamination, disposal of human and chicken feces, water and food storage.
Change in availability and accessibility of safe water storage containers, hygienic toilet, handwashing station, child potty (for >6 months to 2 year old children), and covers for cooked food. | Baseline and 12 months after intervention; ~5 min/assessment
  This will be measured with self-reported behaviors, as well as observations of water storage facilities, latrine quality, handwashing station and child potty.
Change in responsive feeding and interactions during mealtime | Baseline and 12 months after intervention; ~5 min/assessment
  This will be assessed with self-reported interactions mother/caregiver follow during feeding (complementary foods) to their 6-24 months old children

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Luby, Dr., Principal Investigator — Stanford University
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Derived] Sultana J, Pitchik HO, Shoab AK, Huda TMN, Hasan R, Akter F, Jahir T, Khobair Hossain M, Das JB, Amin MR, Yeasmin F, Khan R, Forsyth JE, Kwong LH, Rashid J, Ashrafee S, Rahman M, Mridha MK, Tofail F, Winch PJ, Luby SP, Fernald LCH. Evaluation of a multicomponent child development intervention delivered through the government health system: a feasibility study. BMJ Glob Health. 2025 Jul 20;10(7):e018736. doi: 10.1136/bmjgh-2024-018736. PMID 40685160
- [Derived] Winters S, Pitchik HO, Akter F, Yeasmin F, Jahir T, Huda TMN, Rahman M, Winch PJ, Luby SP, Fernald LCH. How does women's empowerment relate to antenatal care attendance? A cross-sectional analysis among rural women in Bangladesh. BMC Pregnancy Childbirth. 2023 Jun 13;23(1):436. doi: 10.1186/s12884-023-05737-9. PMID 37312017